CLINICAL TRIAL: NCT02851576
Title: Generation of Clinical Grade Adenovirus Specific T Cells for Adoptive Immunotherapy After Allogeneic Stem Cell Transplantation : Clinical Trial
Brief Title: Clinical Grade Adenovirus Specific T Cells for Immunotherapy After Allogeneic Stem Cell Transplantation (CTL-ADV)
Acronym: CTL-ADV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A01029-30
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Adenovirus Infection
Keywords: Adenovirus
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infusion of ADV specific T cells (Experimental): This one arm study consists in ADV-specific T cell infusion after HSCT from a (M)MUD or, for the first time, from a haploidentical donor for patients having undergone previous UCB transplantation, in the event of refractory ADV infection or disease. Specific anti-ADV immune reconstitution was observed in all patients, and viral load clearance in all but one.
  Interventions: Other: Infusion of ADV specific T cells

INTERVENTIONS:
Other: Infusion of ADV specific T cells — Cell engineering

SUMMARY:
Fourteen patients will be included for infusion of adenovirus-specific T-cells generated by a clinical grade IFN-γ based immunomagnetic isolation from a leukapheresis from their original donor or a haploidentical donor, in case of Umbilical cord blood transplantation, in the event of refractory ADV infection or disease.

DETAILED DESCRIPTION:
Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) has improved over the last decades. However, after HSCT and especially with matched unrelated, cord blood or haploidentical donors, patients often experience a deep immunodeficiency, increasing susceptibility to viral infections. Among them, adenovirus (ADV) systemic infection, often refractory to antiviral treatment, is associated with a high mortality rate up to 50% (even more in children). Viremia monitoring after HSCT has contributed to improve survival allowing the implementation of a pre-emptive anti-viral treatment before any appearance of clinical signs of ADV disease. Nevertheless, no anti-viral drug is authorized for ADV infections, although intravenous (IV) cidofovir seemed to be, up to now, the most efficient. However, nephrotoxicity, especially tubular dysfunction, is often described, requiring hydratation and uroprotection with probenecid and limiting the treatment period.

Meanwhile, adoptive transfer of ADV-specific T cells, prepared with an immunomagnetic clinical grade technology, is becoming an alternative treatment that has already proved feasible, safe and helpful in viral clearance and immune reconstitution related to an in vivo expansion of ADV-specific T cells leading to clinical improvement (Feuchtinger et al, 2006, 2015; Qazim et al, 2013). Our team proposes a multicenter Phase I/II clinical trial with ADV-specific T cells where 14 patients, with refractory ADV infection or disease after unrelated Peripheral blood or umbilical cord blood HSCT, are included.

ELIGIBILITY:
Inclusion Criteria:

* Study Population : adults or children
* Allogeneic hematopoietic stem cell (bone marrow and peripheral blood stem cell, umbilical cord blood (UCB))
* sibling or matched unrelated donors 10/10 or 9/10 ((M)MUD) or haploidentical donor in case of UCB transplantation

Within 18 months after HSCT, occurrence of:

- An adenovirus infection without clinical symptoms (except fever with unknown origin) definitively due to this infection, after treatment failure during at least 2 weeks with Cidofovir (5 mg/kg/week).

To determine ADV infection, 2 consecutive viremia performed at 4 days interval must be higher than viral threshold of 500 copies/mL (with significant increase between these 2 analysis and at least 0, 5 log when the first viremia is equal to 500 cp/mL).

* Probable or definitive adenovirus infection after Cidofovir treatment failure, 5 mg/kg/week (according to Wisconsin's criteria)
* and/or renal toxicity or major intolerance to anti-viral drug
* and/or in case Cidofovir is not available in France
* Acute or Chronic GVHD with acute form grade II or less, controlled after 2 lines of treatment at the most.

Or controlled Chronic GVHD

- Life expectancy > 1 month at the time of inclusion

Exclusion Criteria:

* Graft failure
* Derogatory HSCT
* Acute or Chronic GVHD in acute form with grade > II, uncontrolled after 2 lines of immunosuppressive agents.
* Patients with grade > III clinical or biological toxicities (according to OMS classification)
* Chronic GVHD uncontrolled
* Immediate life-threatening
* Patients have not signed informed consent

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Graft Versus Hot Disease (GVHD) grade >2 | 1 month
  No occurrence of acute Graft Versus Hot Disease (GVHD) grade >2 and/or extensive chronic GVHD and no reactivation or worsening of acute or chronic GVHD during the first month following infusion.

SECONDARY OUTCOMES:
Follow-up of ADV viral load | 90 days
  Follow-up of ADV viral load by quantitative Polymerase Chain Reaction (PCR) : Decrease > 0.5 Log
Follow-up of anti-ADV immune response | 90 days
  Follow-up of anti-ADV immune response in the recipient (developing a specific immune response based on in vivo CTL expansion evaluated by IFN ELISPOT or intracellular cytokine staining).

CONTACTS AND LOCATIONS:
Overall Officials: Cécile POCHON, Doctor, Principal Investigator — Central Hospital, Nancy, France; Laurence CLEMENT, Doctor, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Hospitalier Universitaire de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aissi-Rothe L, Decot V, Venard V, Jeulin H, Salmon A, Clement L, Kennel A, Mathieu C, Dalle JH, Rauser G, Cambouris C, de Carvalho M, Stoltz JF, Bordigoni P, Bensoussan D. Rapid generation of full clinical-grade human antiadenovirus cytotoxic T cells for adoptive immunotherapy. J Immunother. 2010 May;33(4):414-24. doi: 10.1097/CJI.0b013e3181cc263b. PMID 20386465
- [Background] Feucht J, Opherk K, Lang P, Kayser S, Hartl L, Bethge W, Matthes-Martin S, Bader P, Albert MH, Maecker-Kolhoff B, Greil J, Einsele H, Schlegel PG, Schuster FR, Kremens B, Rossig C, Gruhn B, Handgretinger R, Feuchtinger T. Adoptive T-cell therapy with hexon-specific Th1 cells as a treatment of refractory adenovirus infection after HSCT. Blood. 2015 Mar 19;125(12):1986-94. doi: 10.1182/blood-2014-06-573725. Epub 2015 Jan 23. PMID 25617426
- [Background] Feuchtinger T, Matthes-Martin S, Richard C, Lion T, Fuhrer M, Hamprecht K, Handgretinger R, Peters C, Schuster FR, Beck R, Schumm M, Lotfi R, Jahn G, Lang P. Safe adoptive transfer of virus-specific T-cell immunity for the treatment of systemic adenovirus infection after allogeneic stem cell transplantation. Br J Haematol. 2006 Jul;134(1):64-76. doi: 10.1111/j.1365-2141.2006.06108.x. PMID 16803570
- [Derived] Qian C, Campidelli A, Wang Y, Cai H, Venard V, Jeulin H, Dalle JH, Pochon C, D'aveni M, Bruno B, Paillard C, Vigouroux S, Jubert C, Ceballos P, Marie-Cardine A, Galambrun C, Cholle C, Clerc Urmes I, Petitpain N, De Carvalho Bittencourt M, Decot V, Reppel L, Salmon A, Clement L, Bensoussan D. Curative or pre-emptive adenovirus-specific T cell transfer from matched unrelated or third party haploidentical donors after HSCT, including UCB transplantations: a successful phase I/II multicenter clinical trial. J Hematol Oncol. 2017 May 8;10(1):102. doi: 10.1186/s13045-017-0469-0. PMID 28482908